CLINICAL TRIAL: NCT01838642
Title: A Phase II Study of Ponatinib in Advanced or Metastatic Medullary Thyroid Cancer
Brief Title: Ponatinib for Advanced Medullary Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruiting halted prematurely and will not resume. New study to open soon.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130108; 13-C-0108
Record Dates: First submitted 2013-04-20; First posted 2013-04-24 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Thyroid Neoplasms
Keywords: Monoclonal Antibody; AP24534; RET Mutation Positive; RET Mutation Negative; RET Inhibitor
MeSH Terms: conditions — Thyroid Neoplasms | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RET mutation positive participants (Active Comparator): Rearranged during transfection (RET) mutation positive
  Interventions: Drug: Ponatinib
- RET mutation negative participants (Active Comparator): Rearranged during transfection (RET) mutation negative
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib tablets will be administered orally, continually, once daily at a dose of 30 mg. A cycle of ponatinib is defined as 28 consecutive days starting with the first day of the treatment cycle. Treatment will be administered primarily in an outpatient setting.

SUMMARY:
Background:

* Medullary thyroid cancer (MTC) represents 5% of thyroid cancers and presents as a hereditary (25% of cases) or sporadic (75% of cases) neuroendocrine malignancy.
* MTC arises from the parafollicular C-cells of the thyroid.
* Germline mutations in the rearranged during transfection (RET) proto-oncogene occur in virtually all of hereditary MTC cases, and somatic RET mutations occur in 50% of sporadic cases.
* Drugs targeting RET kinase such as vandetanib and cabozantinib have shown efficacy in the treatment of advanced or metastatic MTC, however, more effective RET inhibitors are needed for previously untreated patients as well as patients who have become refractory to other molecular targeted therapeutics (MTTs).
* Ponatinib, a drug that is Food and Drug Administration (FDA) approved as a therapy for chronic myelogenous leukemia

(CML) and Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL), is a potent inhibitor of RET kinase.

Primary Objective:

-To determine the objective overall response rate (complete response [CR] + partial response

[PR] by Response Evaluation Criteria in Solid Tumors (RECIST) to ponatinib in the treatment of patients with advanced or metastatic MTC previously treated with cabozantinib and vandetanib who: 1) have tumors with RET mutations and 2) have tumors without RET mutations.

Eligibility:

* Patients must have histologically confirmed, unresectable, locally advanced or metastatic MTC, with measurable disease by RECIST criteria.
* Patients must have disease amenable to biopsy and be willing to undergo biopsy for molecular analysis, and also have adequate archival material from their thyroidectomy or from a tumor biopsy obtained prior to beginning any systemic therapy.
* Patients must have failed or been intolerant to prior treatment with both cabozantinib and vandetanib.
* The last dose of prior systemic therapy must be more than 28 days prior to the first dose of ponatinib
* Radiation therapy is permitted if the last treatment was received more than 28 days prior to the first dose of ponatinib.

Design:

* Open label phase II trial with 2 treatment groups:
* RET mutation positive MTC, previously treated with vandetanib and cabozantinib
* RET mutation negative MTC, previously treated with vandetanib and cabozantinib
* Patients will receive ponatinib 30 mg orally daily until disease progression or until the development of intolerable side effects.
* Tumor response will be assessed by RECIST 1.1 criteria at 8 weeks and then every 12 weeks thereafter. After one year on study, tumor response will be assessed every 16 weeks.
* Patients will have a biopsy of their MTC for molecular analysis prior to initiating treatment with ponatinib. Patients will also have a biopsy of their MTC at the time of tumor progression, should that occur.

DETAILED DESCRIPTION:
Background:

* Medullary thyroid cancer (MTC) represents 5% of thyroid cancers and presents as a hereditary (25% of cases) or sporadic (75% of cases) neuroendocrine malignancy.
* MTC arises from the parafollicular C-cells of the thyroid.
* Germline mutations in the rearranged during transfection (RET) proto-oncogene occur in virtually all of hereditary MTC cases, and somatic RET mutations occur in 50% of sporadic cases.
* Drugs targeting RET kinase such as vandetanib and cabozantinib have shown efficacy in the treatment of advanced or metastatic MTC, however, more effective RET inhibitors are needed for previously untreated patients as well as patients who have become refractory to other molecular targeted therapeutics (MTTs).
* Ponatinib, a drug that is Food and Drug Administration (FDA) approved as a therapy for chronic myelogenous leukemia

(CML) and Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL), is a potent inhibitor of RET kinase.

Primary Objective:

-To determine the objective overall response rate (complete response [CR] + partial response [PR] by Response Evaluation Criteria in Solid Tumors (RECIST) to ponatinib in the treatment of patients with advanced or metastatic MTC previously treated cabozantinib and vandetanib who: 1) have tumors with RET mutations and 2) have tumors without RET mutations.

Eligibility:

* Patients must have histologically confirmed, unresectable, locally advanced or metastatic MTC, with measurable disease by RECIST criteria.
* Patients must have disease amenable to biopsy and be willing to undergo biopsy for molecular analysis, and also have adequate archival material from their thyroidectomy or from a tumor biopsy obtained prior to beginning any systemic therapy.
* Patients must have failed or been intolerant to prior treatment with both cabozantinib and vandetanib.
* The last dose of prior systemic therapy must be more than 28 days prior to the first dose of ponatinib.
* Radiation therapy is permitted if the last treatment was received more than 28 days prior to the first dose of ponatinib.

Design:

* Open label phase II trial with 2 treatment groups:
* RET mutation positive MTC, previously treated with vandetanib and cabozantinib
* RET mutation negative MTC, previously treated with vandetanib and cabozantinib
* Patients will receive ponatinib 30 mg orally daily until disease progression or until the development of intolerable side effects.
* Tumor response will be assessed by RECIST 1.1 criteria at 8 weeks and then every 12 weeks thereafter. After one year on study, tumor response will be assessed every 16 weeks.
* Patients will have a biopsy of their MTC for molecular analysis prior to initiating treatment with ponatinib. Patients will also have a biopsy of their MTC at the time of tumor progression, should that occur.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of localized or metastatic unresectable medullary thyroid cancer (MTC). The histological diagnosis of MTC must be confirmed on review of submitted tumor tissue by the Laboratory of Pathology in the National Cancer Institute
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan.
* Disease amenable to biopsy and agree to undergo biopsy for molecular analysis
* The last dose of previous therapy targeting rearranged during transfection (RET) kinase must be given at least 4 weeks prior to the first dose of ponatinib.
* Previous treatment with cytotoxic chemotherapy, immunotherapy, or radiotherapy are permitted, if the last dose was given at least 4 weeks prior to the first dose of ponatinib
* Patient must have failed (progressed on or been intolerant of) prior treatment with cabozantinib and vandetanib.
* Age greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Normal organ and marrow function as defined below:

  * Leukocytes greater than or equal to microL
  * Absolute neutrophil count 1,500/microL
  * Platelet count greater than or equal to 100,000 microL
  * Total bilirubin < 1.5 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase(SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) < 2.5 times institutional ULN or < 5 times ULN if liver involvement
  * Prothrombin Time < 1.5 times ULN
  * Creatinine < 1.5 times ULN
  * Lipase less than or equal to 1.5 times ULN
* Negative pregnancy test for women of childbearing potential. The effects of ponatinib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Normal QT interval corrected (Fridericia) (QTcF) on screening electrocardiogram (ECG) evaluation, defined as QTcF of less than or equal to 450 ms in males or less than or equal to 470 ms in females.
* Ability to understand and the willingness to sign a written informed consent document and follow the guidelines of the clinical protocol including visits to National Cancer Institute (NCI), Bethesda, Maryland for treatment and follow up visits.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agent.
* Patients with brain metastases or spinal cord compression unless they completed radiation therapy greater than or equal to 4 weeks prior to the first dose of ponatinib and are stable without steroids or anti-convulsant therapy for greater than or equal to 10 days.
* Medications that are known to be associated with Torsades de Pointes.
* Uncontrolled hypertension (systolic blood pressure > 150 or diastolic blood pressure > 100
* Significant or active cardiovascular disease, specifically including but not restricted to:

  * History of myocardial infarction
  * History of atrial or ventricular arrhythmia
  * Unstable angina within 6 months prior to first dose of ponatinib
  * History of congestive heart failure
  * Left ventricular ejection fraction fraction (LVEF) less than lower limit of normal
  * History of peripheral arterial occlusive disease
  * History of cerebrovascular accident or transient ischemic attack
  * Venous thromboembolism including deep venous thrombosis or pulmonary embolism within 6 months prior to enrollment
* A history of pancreatitis or alcohol abuse
* Uncontrolled hypertriglyceridemia (> 450 mg/dL)
* Major surgery (with the exception of minor surgical procedures, such as catheter placement or tumor biopsy) within 28 days prior to the first dose of ponatinib
* Ongoing or active infection including known history of human immunodeficiency virus [HIV], hepatitis B virus [HBV], or hepatitis C virus[HCV]. Testing for these viruses is not required in the absence of a history of infection.
* Suffer from any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of the safety of the study drug
* Evidence of a bleeding diathesis that cannot be corrected with standard therapy or factor replacement
* Presence of another primary malignancy within the past 2 years (except for nonmelanoma skin cancer or cervical cancer in situ. Prior prostate cancer is also permitted if prostatic specific antigen (PSA) is now undetectable.)
* Pregnant or lactating

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lakhani VT, You YN, Wells SA. The multiple endocrine neoplasia syndromes. Annu Rev Med. 2007;58:253-65. doi: 10.1146/annurev.med.58.100305.115303. PMID 17037976
- [Background] Modigliani E, Cohen R, Campos JM, Conte-Devolx B, Maes B, Boneu A, Schlumberger M, Bigorgne JC, Dumontier P, Leclerc L, Corcuff B, Guilhem I. Prognostic factors for survival and for biochemical cure in medullary thyroid carcinoma: results in 899 patients. The GETC Study Group. Groupe d'etude des tumeurs a calcitonine. Clin Endocrinol (Oxf). 1998 Mar;48(3):265-73. doi: 10.1046/j.1365-2265.1998.00392.x. PMID 9578814
- [Background] Moley JF, DeBenedetti MK. Patterns of nodal metastases in palpable medullary thyroid carcinoma: recommendations for extent of node dissection. Ann Surg. 1999 Jun;229(6):880-7; discussion 887-8. doi: 10.1097/00000658-199906000-00016. PMID 10363903
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-C-0108.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in the RET mutation negative group; study closed prematurely.
Groups:
- RET Mutation Positive Participants.: Rearranged during transfection (RET)
  Ponatinib: Ponatinib tablets will be administered orally, continually, once daily at a dose of 30 mg. A cycle of ponatinib is defined as 28 consecutive days starting with the first day of the treatment cycle. Treatment will be administered primarily in an outpatient setting.
Period: Overall Study
Arm/Group | RET Mutation Positive Participants.
Started | 3
Completed | 2
Not Completed | 1
Not completed — Died on study | 1

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the RET mutation negative group; study closed prematurely.
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.13 (5.83)
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate.
Description: Defined as the percentage of participants with a best response (complete response (CR) + partial response (PR)) recorded from the start of the treatment until disease progression/recurrence assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is the disappearance of all target lesions. Any pathological lymph nodes (Whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 2-4 months
Population: No participants were enrolled in the RET mutation negative group; study closed prematurely.
Measure: Number; unit: percentage of participants
Groups:
- RET Mutation Positive Participants: Rearranged during transfection) (RET)
  Ponatinib: Ponatinib tablets will be administered orally, continually, once daily at a dose of 30 mg. A cycle of ponatinib is defined as 28 consecutive days starting with the first day of the treatment cycle. Treatment will be administered primarily in an outpatient setting.
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 3
percentage of participants
  Complete Response | 0
  Partial Response | 0

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: 2-4 months
Population: No participants were enrolled in the RET mutation negative group; study closed prematurely.
Measure: Mean (Full Range); unit: months
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 3
months | 3.01 [2.07 to 4.13]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 17 months and 19 days
Population: No participants were enrolled in the RET mutation negative group; study closed prematurely.
Measure: Number; unit: participants
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 3
participants | 3

4. Secondary Outcome: Molecular Differences in Advanced Medullary Thyroid Cancer (MTC)
Description: Compare the molecular profile of tumor deoxyribonucleic acid (DNA) prior to treatment with the molecular profile at the time of progression. Prior to the first dose of ponatinib and at time of progression, subjects were to undergo a biopsy of the primary tumor or any metastatic site for analysis of tumor DNA for rearranged during transfection (RET) or rat sarcoma (RAS) mutation. Progression is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% decrease in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Prior to the first dose of ponatinib
Population: Although molecular profiling was to be completed prior to first dose of ponatinib and at time of progression, samples were tested on arrival only as mutational status was an eligibility requirement. No participants were enrolled in the RET mutation negative group; study closed prematurely.
Measure: Number; unit: participants
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 3
participants
  RET mutation | 3
  RAS mutation | 0

5. Secondary Outcome: Changes in Serum Levels of MTC Tumor Markers Calcitonin (CTN) and Its Relation With Clinical Response
Description: Responders are those subjects with a best biomarker response of complete response (CR) or partial response (PR) and who achieve a clinical response of CR or PR assessed by the following criteria. Biomarker: complete response (CR) is normalization (</= upper limit of normal (ULN)) of CTN (i.e., normal <10 pg/mL) following treatment, confirmed with a repeat CTN level at least 4 weeks apart. Partial response (PR) is a >/=50% decrease in the CTN level relative to baseline level, confirmed with a repeat CTN level at least 4 weeks apart. Clinical: complete response (CR) is an average of 0-2 formed stools per day for a period of at least 4 weeks. Partial response (PR) is a >50% decrease in the average stool frequency relative to baseline and a change in stool consistency from watery to loose (partially formed) for a period of at least 4 weeks.
Time Frame: Baseline to 4 weeks
Population: None of the participants achieved a clinical response and no data were collected for this assessment. No participants were enrolled in the RET mutation negative group; study closed prematurely.
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Objective Response to Ponatinib
Description: Objective response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is the disappearance of all target lesions. Any pathological lymph nodes (Whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. Stable disease (SD) is neither shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: up to 4 cycles of treatment with ponatinib
Population: One participant died on study during cycle 2. No participants were enrolled in the RET mutation negative group; study closed prematurely.
Measure: Number; unit: participants
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 2
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Progressive Disease (PD) | 2
  Stable Disease (SD) | 0

7. Secondary Outcome: Changes in Serum Levels of MTC Tumor Markers Carcinoemybryonic Antigen (CEA) and Its Relation With Clinical Response
Description: Responders are those subjects with a best biomarker response of complete response (CR) or partial response (PR) and who achieve a clinical response of CR or PR assessed by the following criteria. Biomarker: complete response (CR) is normalization (</= upper limit of normal (ULN)) of CTN (i.e., normal 0-2.5 mcg/L) following treatment, confirmed with a repeat CEA level at least 4 weeks apart. Partial response (PR) is a >/=50% decrease in the CEA level relative to baseline level, confirmed with a repeat CEA level at least 4 weeks apart. Clinical: complete response (CR) is an average of 0-2 formed stools per day for a period of at least 4 weeks. Partial response (PR) is a >50% decrease in the average stool frequency relative to baseline and a change in stool consistency from watery to loose (partially formed) for a period of at least 4 weeks.
Time Frame: Baseline to 4 weeks
Population: as for outcome 5
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time between the first day of treatment to the day of disease progression.
Time Frame: up to 6 months
Population: No participants were enrolled in the RET mutation negative group; study closed prematurely.
Measure: Mean (Full Range); unit: months
Arm/Group | RET Mutation Positive Participants
Number analyzed (Participants) | 3
months | 4.7 [2.1 to 6]

ADVERSE EVENTS:
Time Frame: 17 months and 19 days
Description: No participants were enrolled in the RET mutation negative group; study closed prematurely.
Arm/Group | RET Mutation Positive Participants
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RET Mutation Positive Participants (N=3)
Death NOS (General disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RET Mutation Positive Participants (N=3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Chills (General disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Fatigue (General disorders) | 2 (3)
Fever (General disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lipase increased (Investigations) | 3 (3)
Localized edema (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No